CLINICAL TRIAL: NCT05536713
Title: Understanding Patient Preference on Colorectal Cancer Screening Options
Acronym: U-Screen
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Karen Kim, Professor Department of Medicine, Milton S. Hershey Medical Center
Other Study IDs: IRB22-0345
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Federally Qualified Health Center 1: Patients who received an order for colorectal cancer screening, either using a stool-based test or colonoscopy, but failed to complete the screening after six months will be recruited to participate in the study.
  Interventions: Device: Guardant SHIELD blood-based colorectal cancer screening test
- Federally Qualified Health Center 2: Patients who received an order for colorectal cancer screening, either using a stool-based test or colonoscopy, but failed to complete the screening after six months will be recruited to participate in the study.
  Interventions: Device: Guardant SHIELD blood-based colorectal cancer screening test
- Federally Qualified Health Center 3: Patients who received an order for colorectal cancer screening, either using a stool-based test or colonoscopy, but failed to complete the screening after six months will be recruited to participate in the study.
  Interventions: Device: Guardant SHIELD blood-based colorectal cancer screening test

INTERVENTIONS:
Device: Guardant SHIELD blood-based colorectal cancer screening test — The Guardant SHIELD test combines a next-generation sequencing (NGS) based assay and a protein assay for the qualitative detection of colorectal cancer-derived tumor signal in the blood of patients at average risk for CRC. The Guardant SHIELD was developed at Guardant Health's clinical laboratory, a certified laboratory under the Clinical Laboratory Improvement Amendments of 1988 (CLIA), to perform high-complexity clinical laboratory testing. The test has not been cleared or approved by the U.S. Food and Drug Administration (FDA); however, its performance has been established through a clinical trial, the ECLIPSE study (ClinicalTrials.gov Identifier: NCT04136002). The ECLIPSE clinical trial was a prospective, multi-site registration study and reached the targeted enrollment of 12,750 patients in December 2021.

SUMMARY:
Early detection by screening significantly reduces mortality from colorectal cancer (CRC). However, CRC screening rates have plateaued, with a considerable segment of the population remaining unscreened. Not being up to date with screening was associated with an approximate 3-fold risk for CRC-related mortality. There are different well-established CRC screening modalities, including invasive and non-invasive, which detect both polyps and cancer or cancer alone. Colonoscopy remains the dominant screening modality in the U.S.; however, colonoscopy uptake is low due to the invasiveness, perception of discomfort and embarrassment, logistical challenges, cost, and potential risks.

Increasing patient compliance and adherence to screening is critical to improving CRC outcomes. A key to enhancing screening participation is patient acceptance of the testing method. A blood-based screening test presents an opportunity to overcome some challenging barriers. Blood-based tests are non-invasive compared to colonoscopy and can easily be part of a standard medical office appointment for a wellness check or scheduled visits to manage chronic illnesses and be completed at the point of care. This study will examine patient preference to use a blood-based screening test and compliance with CRC screening recommendations after failing to complete the FIT (Fecal Immunochemical Test)/FOBT (Fecal Occult Blood Test) or colonoscopy order in six months. Compliance with CRC screening is particularly poor among medically underserved populations, and most of these vulnerable individuals use federally qualified health centers (FQHCs) to obtain care. Implementing a blood-based screening test at FQHCs has the potential to improve CRC screening uptake and adherence and improve health disparities in medically underserved populations.

This study seeks to answer the following four questions: 1) What is the acceptability of a blood-based screening as an alternative for patients who failed to complete a prior order using traditional screening methods? 2) Are patients who failed to comply with traditional screening methods more likely to comply with a blood-based screening test? 3) What is the effect of offering a blood-based screening test for patients who are non-compliance with traditional screening methods on overall CRC screening rates? 4) What are the facilitators and barriers to implementing the blood-based screening test in clinical settings?

DETAILED DESCRIPTION:
Significance

A key to improving screening participation is patient acceptance of the testing method. Indeed, all screening modalities have benefits over time, and compliance with testing is essential for successful screening. A blood-based screening test can easily be part of a routine clinic visit, and the patient can complete the test while still at the clinic. Patients are accustomed to providing blood samples for other screening tests, such as cholesterol screening (the national screening rate was 87% in 2019), and the use of a blood-based CRC screening test is more in line with a patient's expectations of medical care. On January 19, 2021, the Centers for Medicare and Medicaid Services announced that the blood-based biomarker test is an appropriate CRC screening once every three years for Medicare patients when performed in a CLIA-certified laboratory, ordered by a treating physician, and the blood-based biomarker screening test has a sensitivity greater than or equal to 74% and a specificity greater than or equal to 90% in the detection of CRC.

The last decades have seen many discovery studies identifying promising biomarkers of CRC. Improving testing methods for blood-based CRC testing have been developed and implemented in clinical settings as well. The first blood-based CRC screening test, SEPT9 DNA (Epi proColon), was approved by the FDA in 2016 for persons at average risk for CRC who have chosen not to undergo screening by existing guideline-recommended methods. This study will offer a lab-developed Guardant SHIELD blood-based CRC screening test to patients who failed to complete a stool-based screening test or a colonoscopy six months after receiving an order from their providers. The Guardant SHIELD blood-based screening test will be free to the patients with an order from their providers. The Guardant SHIELD test is a multimodal blood-based colorectal neoplasia detection assay incorporating ctDNA (circulating tumor DNA) assessment of somatic mutations and tumor-derived methylation and fragmentomic patterns to maximize early-stage CRC detection sensitivity. Overall, the Guardant SHIELD blood-based test has a CRC sensitivity of 91% and a specificity of 94%, meeting the Centers for Medicare and Medicaid Services requirement (74% for sensitivity and 90% for specificity). All the blood samples collected in this study will be processed at the CLIA-certified Guardant Health Laboratory.

Compliance by age-eligible patients is essential to the success of any screening program. However, the acceptance by health care providers and the health care system is also critical, and especially colonoscopy remains the dominant modality for CRC in the U.S. Applying the current state of research evidence to health care involves fostering the adoption, implementation, spread, and sustainability of new evidence-based interventions to care. Furthermore, transferring effective interventions into real-world settings and maintaining them is a complicated, long-term process that requires complex phases of intervention diffusion. In this study, the investigators will examine the inclusion of a blood-based screening option to increase patient compliance with CRC screening while developing implementation strategies to facilitate the adoption of a new blood-based screening test at primary care clinics.

The overall goal of the study is two-fold: 1) examine patient preference when a blood-based CRC screening option is available, and compliance with CRC screening, especially among diverse and vulnerable populations; and 2) understand how to increase the adoption, implementation, and sustainability of an evidence-based screening method to improve CRC screening uptake and adherence.

Study Design

This study will use an Effectiveness-Implementation (Hybrid Type II) Design to examine patient preference and screening compliance when a blood-based test screening option is available and our implementation strategies simultaneously. The Hybrid Type II Design provides rapid translational gains, practical implementation strategies, and helpful information for decision-makers. The stepped wedge cluster randomized trial will be used to examine the blood-based test option in improving screening acceptance and compliance. The stepped wedge is a pragmatic study design and retains some randomization elements as a controlled trial. The stepped wedge design includes an initial period of no exposure. Then one group (or group of clusters) will be randomized to cross from the control to the intervention. All groups will be exposed to the intervention component but not at the same time. Each group contributes to exposed and unexposed observations and acts as its control. In addition, if every cluster shows similar change after crossing to the intervention condition and does not change at other times, it will provide compelling evidence that the change resulted from the intervention even with a limited number of clusters. Furthermore, the feature of multiple data collection points in stepped wedge design allows the researcher to capture the impact of an intervention when such impact develops over time or when the intervention needs an initial adjustment period before becoming embedded in the settings. This feature is valuable for this project when the diffusion of innovation takes time. In this project, the investigators will first implement the blood-based screening test at one of the FQHCs. After three months, the investigators will implement the same intervention at the second FQHC and three months later at the third FQHC.

Study Sites

The investigators will implement the blood-based screening test at three FQHCs, two in Illinois and one in Indiana. Each FQHC has a cluster of 10 to 17 primary care clinics.

Study Procedures

1. Recruitment

   The investigators will collaborate with the patient navigator at partner sites to identify patients who failed to complete their screening after six months. The patient navigator will share study recruitment flyers with the identified patients. If the patient is interested in the blood-based screening test, the navigator will refer them to the study coordinator. The study coordinator will provide patient education on the Guardant SHIELD blood-based screening test, answer questions, and mail education material to the patient when requested.
2. Informed Consent and Enrollment

   Participants who provide informed consent, meet the eligibility criteria, and give a blood sample for CRC screening will be enrolled. Participants will have their blood drawn during their next clinic visit after signing the consent form. A phlebotomist at the clinic will draw the blood and send it to the Guardant Health Laboratory for testing vid FedEx.
3. Screening Result and Follow-up Guardant Health Laboratory will share the test result with the ordering provider. Ordering providers will discuss the test finding with their patients and refer patients to follow-up colonoscopy in the case of a positive test result. Before the implementation, providers at our partner FQHCs will attend a training session delivered by Guardant Health scientists on the Guardant SHIELD blood-based screening test, including interpreting the results. If a study participant receives a positive result, the patient navigator at our partner sites and our study coordinator will assist with colonoscopy scheduling and educate on bowel preparation. The investigators will work with Guardant Health to support uninsured or underinsured patients who have difficulty accessing colonoscopy due to the cost.

Study Endpoints

1. Primary Endpoint

   The primary endpoint is to examine whether the availability of a blood-based screening option, which can be done at the point of service and is familiar to patients, will improve patient compliance with recommended CRC screening. The investigators will assess the effectiveness of the primary endpoint by calculating the number of participants who, otherwise, will not have participated in the CRC screening and completed the Guardant SHIELD blood-based screening test. The investigators will compare the differences within and between health centers and the changes over time. Since the blood-based screening test is a two-step strategy and patients with a positive result must complete a follow-up colonoscopy to maximize the benefit of the screening, the investigators will include colonoscopy referral and completion rates as secondary outcomes during the primary endpoint analysis.
2. Secondary Endpoint

The secondary endpoint analysis is to determine whether the implementation strategies accelerate the adoption and implementation of a blood-based screening test into routine practice. Adoption takes time and is slow at the start, more rapid as adoption increases and then levels off. If the adoption does not reach the critical mass, the process can stall. The adoption rate indicates how fast an idea reaches a certain percentage of people. This study will monitor the adoption rates over time and how long it takes to achieve 2.5%, 16%, and 50% adoption rates (adoption rate = the number of new users / total number of potential users). The investigators will monitor the adoption rate quarterly. In addition, the investigators will also monitor the intensity of use.

Data Collection

During the first three months, The investigators will collect baseline data on non-compliance rates for stool-based tests and colonoscopy. After starting the implementation process, the investigators will collect primary outcome data each quarter until the project's conclusion. At the patient level, the investigators will collect de-identified patient demographic information from EHR, including 1) Health insurance coverage (Yes/No), 2) Race/ethnicity, gender, age, and 3) CRC screening up-to-date status (Yes/No). At the clinic and provider levels, the investigators will collect data on blood-based screening test order rates, blood-based test completion rates, and colorectal cancer screening rates. Since a blood-based screening test is a two-stage strategy and a positive result requires a follow-up colonoscopy, this study will include colonoscopy referral rates, completion rates, and time to colonoscopy completion as secondary outcomes. The investigators will also collect data on patient experiences, including convenience, easiness, and the likelihood of using a blood-based screening test again.

ELIGIBILITY:
Inclusion Criteria:

* Between 45-75 years of age
* Have an average risk for colorectal cancer
* A patient at one of our partner FQHCs
* Received a screening order (either using a stool-based test or colonoscopy) six months ago and failed or refused to complete the screening test
* Able to comprehend and willing to give informed consent
* Able and willing to provide a blood sample per protocol

Exclusion Criteria:

1. Family history

   * One first-degree relative diagnosed with CRC or advanced adenoma at age < 60 years
   * Two first-degree relatives diagnosed with CRC or advanced adenoma at any age
   * Known hereditary gastrointestinal cancer syndromes, such as Lynch Syndrome or Familial Adenomatous and Polyposis (FAP)
2. Personal History

   * History of CRC or adenoma
   * History of cancers
   * History of inflammatory bowel disease, including chronic ulcerative colitis and Crohn's disease
   * Have a recorded up-to-date CRC screening
   * Blood product transfusion in the past 120 days
   * A medical condition that, in the opinion of the patient's health provider, should preclude enrollment in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are age-eligible for colorectal cancer screening based on the U.S. Preventive Service Task Force recommendation guidelines have an average risk for colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Blood-based screening test order rates | 60 days after enrolling in the study
  Number of unique patients who enrolled in the study and received a blood-based screening test order from their providers
Blood-based test compliant rates | 90 days after received an order for a blood-based screening test
  Patients who enrolled in the study , received an order for a blood-based screening test, and completed the test

SECONDARY OUTCOMES:
Follow-up colonoscopy completion rates | 180 days after received the abnormal blood-based screening test result
  Patients who had an abnormal blood-based screening test and completed a follow-up diagnostic colonoscopy
Patient satisfaction with the blood-based test | 30 days after the patient completed the blood-based screening test and received the test result
  Patient is asked to rate their overall experience with the blood-based experience on three domains: convenience, easiness, the likelihood to use the blood-based test again

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kim, MD, Principal Investigator — University of Chicago
Locations (1):
- PCC Community Wellness Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will deposit to Knowledge@Uchicago for open access. Knowledge@UChicago is the University of Chicago's institutional repository.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within 30 days after the manuscript is published.
Access Criteria: Users will complete a user agreement.